CLINICAL TRIAL: NCT02209727
Title: A Phase I Single Dose Escalation Study of 131I-Sibrotuzumab in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Single Dose Escalation Study of 131I-Sibrotuzumab in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1152.6
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- 131I-Sibrotuzumab (Experimental): single therapy dose administered over 60 minutes at week 4
  Interventions: Drug: 131I-Sibrotuzumab

INTERVENTIONS:
Drug: 131I-Sibrotuzumab — 50 mg Sibrotuzumab conjugated with 131I

SUMMARY:
Study to determine the maximum tolerated dose (MTD) and safety profile of a single-dose administration of sibrotuzumab (50 mg) conjugated to an increasing dose of 131 I isotope.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of advanced, non-resectable, and/or metastatic non-small cell lung cancer and at least one previous conventional treatment for advanced disease
* Eastern cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable or evaluable disease, determined by World Health Organization (WHO) criteria using standard imaging modalities, including ultrasound, X-ray, CT and/or Magnetic Resonance Imaging (MRI). Bone scans and/or antibody scans are not to be used to determine the extent of the disease
* Expected survival of ≥ 16 weeks
* At least 18 years of age
* Platelet count ≥ 100 x 10**9/L
* Absolute neutrophil count ≥ 2.0 x 10**9/L
* Aspartate aminotransferase (AST) ≤ 3 x upper limit of normal or < 5 x upper limit of normal if liver metastases are present
* Total bilirubin ≤ 2mg/dL
* Serum creatinine ≤ 2mg/dL
* Ability to provide written informed consent

Exclusion Criteria:

* Known brain metastases
* Exposure to an investigational agent within 30 days prior to receiving the scout dose
* Incomplete recovery from surgery or incomplete healing of an incision site or evidence of infection
* Treatment with cytotoxic chemotherapy, radiation or immunosuppressive therapy within the 30 days (42 days for nitrosoureas and/or mitomycin C) of the scout infusion. Patients using inhaled corticosteroids are considered eligible for enrollment
* Serious illnesses, i.e., active infections requiring antibiotics, bleeding disorders or other serious illnesses precluding the use of either 131I or sibrotuzumab
* Women who are breast-feeding or pregnant
* Men and women who were sexually active and are unwilling to utilize a medically acceptable method of contraception
* Hypertrophic skin disease or autoimmune disease that possibly involves over-expression of fibroblast activation protein (FAP), which can be targeted by the antibody. These diseases include active inflammatory arthritis, cirrhosis, and keloids
* Unstable angina pectoris. Patients prescribed medication to control their angina pectoris must have been on a fixed dose for at least 1 month prior to screening to be eligible for trial enrollment
* Myocardial infarction within 3 months prior to screening
* New York Heart Association (NYHA) Heart failure stage III or IV, or a left ventricular ejection fraction of ≤ 40 %
* Impaired lung function, measured by a decrease in forced expiratory volume at one second (FEV1) to less than 50 % of the predicted normal value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2000-12; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Determination of the dose limiting toxicity (DLT) | up to 12 weeks
Determination of the maximum tolerated dose (MTD) | up to 12 weeks
  MTD is defined as the highest dose below which two patients experience DLT
Occurrence of toxicity | up to 12 weeks
  graded according to the Common Toxicity Criteria (CTC)

SECONDARY OUTCOMES:
Maximum tumor response using the World Health Organisation (WHO) Disease Response Criteria | 8 weeks after therapeutic infusion